CLINICAL TRIAL: NCT06731400
Title: Variability in Human Fatty Acids Profiles Based on Blood Fractions and Metabolic Conditions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Inar Castro Erger, Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 82746224.7.0000.0067
Record Dates: First submitted 2024-11-28; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Atherosclerosis Cardiovascular Disease
Keywords: EPA; DHA; supplementation; leukocytes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EPA Suplementation (Experimental): Six healthy individuals will be supplemented with fish oil for eight weeks, with blood samples collected before and after the intervention.
  Interventions: Dietary Supplement: EPA supplementation

INTERVENTIONS:
Dietary Supplement: EPA supplementation — Six healthy individuals will be supplemented with fish oil contains omega 3 (EPA) for eight weeks, with blood samples collected before and after the intervention.

SUMMARY:
Fatty acids play a crucial role in various metabolic pathways, with their proportions and distributions across different cells and tissues influenced by diet and metabolism. In addition to providing energy through oxidative reactions, fatty acids serve as substrates for the synthesis of numerous molecules involved in cellular signaling processes. Therefore, quantifying fatty acids in biological samples is essential for ensuring the quality of clinical trials involving lipids and for understanding the relationship between fats and health conditions. However, the fatty acid profiles reported in clinical trials can exhibit significant heterogeneity due to both endogenous and exogenous factors, including the metabolic condition of the patients and the specific blood fraction analyzed. This variability makes difficult the comparison of results across studies. Moreover, despite the crucial role of fatty acids in immune response, most results are derived from erythrocytes, plasma, or serum, providing limited information on their variability in leukocytes. Thus, the hypothesis of this study is that metabolic conditions, characterized by fasting or postprandial states, can influence the fatty acid profile depending on the blood fraction analyzed. To evaluate this hypothesis, six healthy individuals will be supplemented with fish oil for eight weeks, with blood samples collected before and after the intervention. Fatty acid levels will be measured using gas chromatography coupled with mass spectrometry in total plasma, phospholipids, erythrocytes, and leukocytes. The results will help estimate the variability caused by metabolic states according to the blood fraction, which is critical when conducting clinical trials in patients where fasting cannot be assured and is essential for comparing fatty acid profiles in studies involving leukocytes.

DETAILED DESCRIPTION:
In summary, it is known that numerous factors can interfere with the effects of administering polyunsaturated fatty acids (n-3 PUFA), including aspects related to the experimental design, such as the form and dosage used, the duration of treatments, the blood fraction and the metabolic state of the individuals. In this context, given the importance of precise quantification of fatty acids in biological samples obtained from humans, the present study will aim to evaluate the variability caused by the administration of fish oil before and after 8 weeks of supplementation. This will involve comparing the fatty acid profiles according to different fractions (plasma, leukocytes, and erythrocytes) and fasting conditions (fasting or post-prandial). In plasma, the analysis will also consider both the total sample and the phospholipidic fraction.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes
* Aged between 20 and 50 years
* No contraindications for the use of fish oil supplements

Exclusion Criteria:

* Use of medications or supplements to reduce triacylglycerols;
* Consumption of fish oil or other supplements/medicines rich in n-3 or n-6 PUFA in the month before the test;
* Consumption of fatty fish (salmon, herring, mackerel, white tuna or sardines) more than twice a month in the month before the test;
* Refusal to avoid PUFA supplements and seafood during the study period;
* Severe heart failure;
* Severe active liver disease;
* Planned coronary intervention or surgery,
* History of acute or chronic pancreatitis;
* Hypersensitivity to fish, shellfish or capsule ingredients;
* Autoimmune diseases requiring immunosuppressive therapy;
* Current corticosteroid use systemic,
* Neoplasms;
* Chemotherapy or radiotherapy within the past 12 months (patients who have undergone curative surgery without requiring additional treatment within the past year may be included);
* Inflammatory bowel disease;
* Chronic diarrhea;
* Significant non-transient hematological abnormalities;
* Kidney dysfunction;
* Severe liver disease;
* Inability to provide informed record;
* Participation in another clinical trial with an experimental agent in the last 90 days;
* Malabsorption syndrome;
* Recent drug or alcohol abuse;
* Atrial fibrillation;
* Bleeding disorders.
* Pregnancy
* Breastfeeding.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-12-03 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
The fasting or postprandial states on the fatty acid profile | From December 2024 to February 2025
  This study will assess whether fasting or postprandial states affect the fatty acid profile based on the blood fraction analyzed. Six healthy individuals will be supplemented with 2 g/day of fish oil for eight weeks, with blood samples collected before and after the intervention. Fatty acid levels will be measured using gas chromatography-mass spectrometry in total plasma, phospholipids, erythrocytes, and leukocytes.
The fasting or postprandial states on the fatty acid profile | From December 2024 to February 2025
  Fatty acid levels will be measured in total plasma, phospholipids, erythrocytes, and leukocytes by fasting or postprandial states.

CONTACTS AND LOCATIONS:
Overall Officials: Inar Castro Erger, Professor, Principal Investigator — Faculty of Pharmaceutical Sciences at the University of São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lozier BK, Kim RN, Zuromski LM, Kish-Trier E, De Biase I, Yuzyuk T. Effect of fasting status and other pre-analytical variables on quantitation of long-chain fatty acids in red blood cells. Prostaglandins Leukot Essent Fatty Acids. 2020 Dec;163:102211. doi: 10.1016/j.plefa.2020.102211. Epub 2020 Nov 19. PMID 33249349
- [Background] BLIGH EG, DYER WJ. A rapid method of total lipid extraction and purification. Can J Biochem Physiol. 1959 Aug;37(8):911-7. doi: 10.1139/o59-099. No abstract available. PMID 13671378
- [Background] Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Ketchum SB, Doyle RT Jr, Juliano RA, Jiao L, Granowitz C, Tardif JC, Ballantyne CM; REDUCE-IT Investigators. Cardiovascular Risk Reduction with Icosapent Ethyl for Hypertriglyceridemia. N Engl J Med. 2019 Jan 3;380(1):11-22. doi: 10.1056/NEJMoa1812792. Epub 2018 Nov 10. PMID 30415628